CLINICAL TRIAL: NCT04287842
Title: Neuroprotective Effect of Desflurane in the Experimental Study: the Impact if Desflurane Preconditioning on the Content of the Phosphorylated Form of GSK-3b in the Neurons of the Rat's Brain in the Model of Ischemia/Reperfusion
Brief Title: Impact if Desflurane Preconditioning on the Content of the Phospho-GSK-3b in the Rat's Neurons in the Model of I/R
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: technical problem
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Des-2014E
Record Dates: First submitted 2015-01-21; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Heart Arrest
Keywords: desflurane; preconditioning
MeSH Terms: conditions — Heart Arrest | interventions — Desflurane; Sevoflurane; Heart Arrest, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- control (No Intervention): Induction of anesthesia: Chloralhydrat intraperitoneal 300 mg/kg. This provides complete suppression of animal responses to pain, fixation, tracheal intubation. After fixation of the animal in the supine position trachea is intubated and mechanic ventlation with air using an animal respirator is performed.
- training ischemia (Experimental): Induction of anesthesia: Chloralhydrat intraperitoneal 300 mg/kg. Comparison of a total GSK-3 and phosphorytated (Ser9) GSK-3beta (pGSK3b) in brain tissuesupracardiac bundle of vessels by means of a special hook after cardiac arrest and absence of ventilation lasts 10 min.
  Interventions: Procedure: Cardiac arrest
- desflurane (Active Comparator): Intervention. Drug: Desflurane. Desflurane 8 vol% anesthesia is introduced. This provides complete suppression of animal responses to pain, fixation, tracheal intubation and cardiac arrest. After fixation of the animal in the supine position trachea is intubated and mechanic ventlation with air using an animal respirator is performed. Surgery: Cardiac arrest is induced by intrathoracic clamping of the supracardiac bundle of vessels by means of a special hook. Period of cardiac arrest and absence of ventilation lasts 10 min. The animal is then resuscitated by means of chest compressions and mechanichal ventilation with air. Cardiac activity and systemic blood circulation recovers within 1 min; spontaneous respiration will be resumed after a period of 4-6 min.
  Interventions: Drug: Desflurane; Procedure: Cardiac arrest
- sevoflurane (Active Comparator): Sevoflurane anesthesia is introduced. This provides complete suppression of animal responses to pain, fixation, tracheal intubation and cardiac arrest. After fixation of the animal in the supine position trachea is intubated and mechanic ventlation with air using an animal respirator is performed. Cardiac arrest is induced by intrathoracic clamping of the supracardiac bundle of vessels by means of a special hook. Period of cardiac arrest and absence of ventilation lasts 10 min. The animal is then resuscitated by means of chest compressions and mechanichal ventilation with air. Cardiac activity and systemic blood circulation recovers within 1 min; spontaneous respiration will be resumed after a period of 4-6 min.
  Interventions: Drug: Sevoflurane; Procedure: Cardiac arrest

INTERVENTIONS:
Drug: Desflurane — Desflurane anesthesia is introduced. This provides complete suppression of animal responses to pain, fixation, tracheal intubation and cardiac arrest.
  Other Names: suprane
  Arms: desflurane
Drug: Sevoflurane — Desflurane anesthesia is introduced. This provides complete suppression of animal responses to pain, fixation, tracheal intubation and cardiac arrest. After fixation of the animal in the supine position trachea is intubated and mechanic ventlation with air using an animal respirator is performed. Cardiac arrest is induced by intrathoracic clamping of the supracardiac bundle of vessels by means of a special hook. Period of cardiac arrest and absence of ventilation lasts 10 min. The animal is then resuscitated by means of chest compressions and mechanichal ventilation with air. Cardiac activity and systemic blood circulation recovers within 1 min; spontaneous respiration will be resumed after a period of 4-6 min.
  Other Names: Sevorane
  Arms: sevoflurane
Procedure: Cardiac arrest — Cardiac arrest is induced by intrathoracic clamping of the supracardiac bundle of vessels by means of a special hook. Period of cardiac arrest and absence of ventilation lasts 10 min. The animal is then resuscitated by means of chest compressions and mechanichal ventilation with air. Cardiac activity and systemic blood circulation recovers within 1 min; spontaneous respiration will be resumed after a period of 4-6 min.
  Arms: desflurane; sevoflurane; training ischemia

SUMMARY:
Endpoint implementation of reactions initiated by ischemia is the mitochondrial transition pore permeability. Mitochondria pores opening results in a release of factors triggering apoptosis primarily the cytochrome С Inhibition of the pores opening protects ischemic damage of the cells. The key enzyme regulating the mitochondrial permeability transition pore is GSK-3b: the phosphorylation of the enzyme inactivates the enzyme and prevents pore opening. Aim of studi is to determine content of the phosphorylatcd GS K-3b in neurons of rat brain in the model of total tschemia/reperfusion.

DETAILED DESCRIPTION:
Endpoint implementation of reactions initiated by ischemia is the mitochondrial transition pore permeability. Mitochondria pores opening results in a release of factors triggering apoptosis. primarily the cytochrome С Inhibition of the pores opening protects ischemic damage of the cells. The key enzyme regulating the mitochondrial permeability transition pore is glycogen synthase-kinase 3b (GSK-3b): the phosphorylation of the enzyme inactivates the enzyme and prevents pore opening. We have shown in previous study that preconditioning with sevoflurane increases the content of the phosphorylated form of 6SK-3b and protects the mitochondria of neurons in rats brain during ischemia/reperfusion. Aim of studi is to determine content of the phosphorylated GS K-3b in neurons of rat brain in the model of total ischemia/reperfusion influenced by: 1 MAC desflurane vs control group; 1 MAC desflurane vs 1 MAC sevoflurane and 1 MAC desflurane vs training ischemia.

ELIGIBILITY:
Inclusion Criteria:

* breeding albino male rats weigh from 180 to 240 g

Exclusion Criteria:

* N/A

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
total GSK-3b and phosphorilated (pGSK-3b) | after 15 minutes of exposition

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, MD,PhD, Principal Investigator — V. Negovskij Reanimatology Research Institute RAMS